CLINICAL TRIAL: NCT00487214
Title: Internet-based, Naturalistic Evaluation of Tolerability and Individual Patient Target Pressures With Bimatoprost 0.03% in Glaucoma
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Other Study IDs: MEDNET2001
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the range of target IOPs set for glaucoma patients starting monotherapy with bimatoprost and to evaluate patient and physician satisfaction with bimatoprost in "real-world" settings

ELIGIBILITY:
Inclusion Criteria:

* Patients with either open-angle glaucoma or ocular hypertension were eligible if they needed bilateral IOP reduction beyond what was achieved with their current medication, or if they were intolerant of other IOP-lowering medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either open-angle glaucoma or ocular hypertension at 41 centers in the United States
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2002-06; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Allergan

REFERENCES:
- See also: (Link to Clinical Trial Results) — http://www.allerganclinicaltrials.com